CLINICAL TRIAL: NCT03501329
Title: Investigation of Change in The WHO-5 Well-Being Index During a Year in a Community Psychiatry in Denmark
Status: Completed | Type: Observational
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Responsible Party: Principal Investigator, Henrik Folker, Principal Investigator (in this area of research), Psychiatric Research Unit, Region Zealand, Denmark
Other Study IDs: UFL-03-18-0170
Record Dates: First submitted 2018-03-21; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Psychiatric Rehabilitation
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Outpatients in Community Psychiatry: Treatment with consultations, social support, psychological and psychopharmacological treatment. This is routine psychiatric care.
  Treatment was not changed as a result of the investigation in itself.
  Interventions: Combination Product: Biological,Psychological and Social support

INTERVENTIONS:
Combination Product: Biological,Psychological and Social support

SUMMARY:
Patient reported quality of life was measured using the WHO-5 Well-Being Index in a group of outpatients in the Community Psychiatry in Holbaek, Denmark.

Methods

The first and last answer were compared and significance of change in various subgroups of patients was estimated using the PSPP statistical program.

DETAILED DESCRIPTION:
Investigation of the change of The WHO-5 Wellbeing Index during a year in a Community Psychiatry in Denmark.

Introduction

In the Community Psychiatry of the town Holbaek part of Region West of The Region Sjaelland in eastern Denmark the WHO-5 Well-Being Index has for 5 years been used in order to obtain the patients personal evaluation of their actual quality of life. That has given the possibility of following changes during the treatment. The questionnaire is easy to understand and to use as part of a consultation. The patients will answer the 5 questions in a few minutes. The WHO-5 questionnaire is thoroughly evaluated internationally and described and used in many clinical situations also outside of psychiatry and fulfill measures of psychometric quality. With this work the intention was to try to answer often critical questions from our administration and from the press and in the society. There was no funding for the work.

ELIGIBILITY:
Inclusion Criteria:

* all patients able and willing to participate

Exclusion Criteria:

* patients with mental conditions making them unable to answer simple questions about their daily life (in general severe psychosis and severe organic mental disorders)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The 752 patients registered as receiving service in district psychiatry during 2017
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in The WHO-5 Well-Being Index | The Time Frame was from the beginning of the participation in the study (baseline) and at the completion of the study participation (approximately 1 year).
  This is a Patient Reported Outcome Measure (PROM) for studying changes in the Well-Being Index during ongoing treatment. In many cases it was not possible to maintain the patients in the study for the intended time period and it was found necessary to accept the latest evaluation as the final measurement of change. It will be possible to report the observation time in months for each single case and to report the median of these periods of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Simonsen, Professor, Study Director — Psykiatrisk Forskningsenhed
Locations (1):
- Psykiatrisk Forskningsenhed, Slagelse, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962